CLINICAL TRIAL: NCT00032279
Title: A Phase II, Multicenter Clinical Trial Evaluating the Use of Humanized Monoclonal Anti-CD3 Antibody Visilizumab(Nuvion) as Second-line Therapy for Glucocorticoid-Refractory, Acute Graft-Versus-Host Disease
Brief Title: Research Study of Visilizumab for Treatment of Glucocorticoid- Refractory Graft Versus Host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Facet Biotech (Industry)
Organization: Facet Biotech (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1589; NCT00042744 (obsolete NCT alias)
Record Dates: First submitted 2002-03-15; First posted 2002-03-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Graft-vs-Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — visilizumab

INTERVENTIONS:
Drug: Visilizumab

SUMMARY:
The purpose of this phase II study is to evaluate an investigational monoclonal antibody for the treatment of glucocorticoid-refractory Graft Versus Host Disease (GVHD). Patients diagnosed with GVHD who have not responded satisfactorily to, or are intolerant of, treatment with standard agents will be considered for entry. Patients will be allowed to continue on their other immunosuppressive drugs at stable doses during the trial. The research is being conducted at up to 20 clinical research sites in the US.

ELIGIBILITY:
* Grade II to IV GVHD
* Clinical findings: skin thickening, joint contraction, oral ulceration, diarrhea.
* History of allogeneic hematopoietic cell transplant (HCT).
* Patients must have failed to respond or clearly progress to previous therapy on or before day +100 posttransplant.
* Patients must have adequate renal, hepatic, cardiac function and hematologic values

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - City of Hope National Medical Center, Duarte, California
  - Stanford University Medical Center, Stanford, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University Hospital, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The New York Hospital Cornell Medical Center, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington